CLINICAL TRIAL: NCT04064398
Title: Evaluation of Gastric Residuals in Preterm Newborns: What Impact Does It Have on Feedings Progression?
Brief Title: Evaluation of Gastric Residuals and Feedings Progression
Acronym: REGAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped when 85% of the sample wascompleted due to the time elapsed and the estimated lack of change in results.
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 190321007
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Infant, Premature, Diseases; Nutrition, Enteral
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine aspiration of gastric residuals (Active Comparator): Infants will have routine aspiration of gastric contents prior to each feeding to monitor the amount of residual gastric contents remaining in the stomach.
  Interventions: Procedure: Aspiration of gastric residuals
- No aspiration of gastric residuals (No Intervention): Infants will not have routine aspiration of gastric contents prior to each feeding.

INTERVENTIONS:
Procedure: Aspiration of gastric residuals — Infants will have routine aspiration of gastric contents prior to each feeding to monitor the amount of residual gastric contents remaining in the stomach.
  Arms: Routine aspiration of gastric residuals

SUMMARY:
This study evaluates the utility of measuring gastric residuals in premature infants born between 26+0 and 33+6 weeks and to determine if its routine use is related with a delay in feedings advancement in this babies compared with no measurement.

DETAILED DESCRIPTION:
The evaluation of gastric residuals as a measure of enteral tolerance in term and especially preterm newborns is a widely used practice in different centers worldwide. However, until now, it continues to be a controversial practice, since its real usefulness is not clear.

Our study proposes to evaluate and compare two groups of preterm newborns born between 26 + 0/7 and 33 + 6/7 weeks, randomized to measure or not measure gastric residuals and determine if this practice delays the full feeding achievement.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 26+0 to 33+6 weeks post-menstrual gestational age.
* Enteral feeds starting during the first week of life.
* Signed informed consent from parents or guardians.

Exclusion Criteria:

* Perinatal asphyxia
* Sepsis and hemodynamic instability
* Major congenital malformations
* Surgical requirement during the first week of life
* Hemodynamic instability and vasoactive drugs requirement
* Moderate or severe respiratory failure with Oxygenation Index > 8

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Time to reach full feeds | Baseline to 8 weeks
  Time in days to reach full feeds defined as receiving 150 ml/kg/day tolerated for at least 24 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina A Salas, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Jorge G Fabres, MD, MSPH, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No